CLINICAL TRIAL: NCT07292532
Title: Out-of-hospital Cardiorespiratory Arrest and Learning Cardiopulmonary Resuscitation in the School Setting: Evidence Synthesis
Brief Title: Learning Cardiopulmonary Resuscitation in the School Setting: RCP-KNOW Project.
Acronym: RCP-KNOW
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Castilla-La Mancha (Other)
Collaborators: Consejería de Educación, Cultura y Deportes de Castilla-La Mancha (Unknown); European Regional Development Fund (Other)
Responsible Party: Principal Investigator, Diana Patricia Pozuelo Carrascosa, Profesora Titular de Universidad, University of Castilla-La Mancha
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SBPLY/23/180225/000060; SBPLY/23/180225/000060 (Other Grant/Funding Number: Junta de Comunidades de Castilla-La Mancha and FEDER Funds)
Record Dates: First submitted 2025-11-14; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-11

CONDITIONS: Healthy Participants; Knowledge Acquisition; Cardiopulmonary Resuscitation (CPR); Children; School

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional CPR teaching (Active Comparator): A 2-hour session of conventional theoretical-practical training with a mannequin, about the BLS sequence to follow in a CPR-OHCA, adapted to the age of schoolchildren, and taught by nursing professionals. Theoretical-practical training on the operation of the semi-automatic defibrillator.
  Interventions: Other: Cardiopulmonary Resuscitation Teaching Intervention in Children
- Video and teaching material (Experimental): A short video (5min) in which the basic sequence of BLS to follow in a CPR-OHCA is explained, accompanied by a puzzle adapted to the age of the children in which the BLS sequence is reflected, but without practice on a mannequin. Theoretical training included in the video about the operation of the semi-automatic defibrillator.
  Interventions: Other: Cardiopulmonary Resuscitation Teaching Intervention in Children

INTERVENTIONS:
Other: Cardiopulmonary Resuscitation Teaching Intervention in Children — Comparation of two type of Cardiopulmonary Resuscitation Teaching Intervention in Children: traditional teaching vs video with puzzle.

SUMMARY:
Title: Out-of-hospital cardiorespiratory arrest and learning cardiopulmonary resuscitation in the school setting: evidence synthesis. CPR-KNOW PROYECT.

Background: The high incidence, associated morbidity and mortality, and the great individual, social and economic impact of out-of-hospital cardiorespiratory arrest (OHCA) make it a priority for all health systems worldwide. To increase the rates of potential first responders who act appropriately, applying basic life support (BLS) measures in the OHCA, the European Resuscitation Council includes among its latest recommendations the training of all school children through the "Kids Save Lives" initiative.

Objectives: to determine, through a randomized clinical trial, the effectiveness of two training strategies for increasing theoretical and practical knowledge of BLS in schoolchildren and adolescents.

Methodology: To evaluate the effectiveness of two (Cardiopulmonary Resuscitation) CPR teaching interventions in improving the following outcome variables: theoretical knowledge and practical skills, CPR quality; as well as its relationship with the anthropometric, sociodemographic and physical condition variables of the schoolers.

* Intervention group 1 (IG1): a 2-hour theoretical-practical session on the BLS sequence taught by a Nursing professional performing the practice with a mannequin. Instructor/school ratio: 1/25 for the theoretical session and a school/mannequin ratio: 2-3/1.
* Intervention group 2 (IG2): a session with short video (approximately 5-10 min) and other teaching resources (puzzle), without practice on a mannequin. Video/school ratio: 1/25 and a school/teaching resource (puzzle) ratio: 1/1.

ELIGIBILITY:
Inclusion Criteria:

* Schools that have at least one complete year of 1st, 2nd, 3rd, 4th, 5th and 6th year of Primary Education, in which the School Council has given its approval for their participation.
* Schoolchildren who wish to participate must:
* Belong to the courses from 1st to 6th grade of Primary Education
* Understand the written and spoken Spanish language
* Not have any physical, mental or cognitive pathology that prevents them from participating in the project.
* Their father/mother or guardian must have signed the informed consent to be able to participate in the project.

Ages: 5 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 550 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Theoretical CPR Knowledge | On the same day as the intervention, before (pre-intervention) and immediately after this (post-intervention) and follow-up (8 months later)
  Theoretical CPR Knowledge measured by a questionnaire.
CPR Practice Skills | On the same day as the intervention immediately after this (post-intervention) and follow-up (8 months later)
  CPR Practice Skills measured with a checklist
Quality of CRP | On the same day as the intervention, immediately after this (post-intervention) and follow-up (8 months later)
  Quality of CPR measured by Little-Anne Mannequin.

OTHER OUTCOMES:
Anthropometry: weight | Immediately post-intervention
  Corporal weight measured in Kilograms
Anthropometry: height | Immediately post-intervention
  Height measured in centimeters
Anthropometry: BMI | Immediately post-intervention
  BMI calculated by the follow form: weight (kg)/height*2 (m)
Anthropometry: corporal composition | Immediately post-intervention
  Percentage of fat mass and percentage of lean mass. Measured by bioimpedance scale Tanita MC-780MA N
Cardiorespiratory fitness | Immediately post-intervention
  Cardiorespiratory fitness measured through Course Navette Test
Muscular strength | Immediately post-intervention
  Muscular strength measured through dynamometry and horizontal jump with feet together
socioeconomic variables | immediately post-intervention
  socioeconomic variables such as: the academic level and economic level of the father and mother

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - CEIP Ciudad Encantada, Cuenca, Cuenca
  - CEIP Isaac Albeniz, Cuenca, Cuenca

IPD SHARING:
Plan to Share IPD: No